CLINICAL TRIAL: NCT02704637
Title: An Evaluation of Non-invasive Acoustic Approach to Detect and Monitor Cerebral Vasospasm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HeadSense Medical (Industry)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-026
Record Dates: First submitted 2016-02-19; First posted 2016-03-10 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2017-02

CONDITIONS: Vasospasm, Intracranial; Subarachnoid Hemorrhage
Keywords: vasospasm
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-1000 recording (Experimental): Each non-invasive recording session with the HS-1000 device will be done for 10 consecutive uninterrupted minutes. Patients will be recorded once daily for the duration of their time in ICU or for up to 14 days total. In the case the PI or a member of the study team positively confirms vasospasm based on clinical assessment or follow-up care during the monitoring period, the patient will be recorded twice daily for up to 14 consecutive days or for their duration in the ICU.
  Interventions: Device: HS-1000

INTERVENTIONS:
Device: HS-1000 — HeadSense (HS)-1000 device, a proprietary non-invasive brain monitor, is expected to safely and accurately monitor physiological signs of the brain with minimal discomfort to patients, providing information about normal or abnormal brain-related conditions and providing decision-making support for physicians

SUMMARY:
HeadSense (HS)-1000 device, a proprietary non-invasive brain monitor, is expected to safely and accurately monitor physiological signs of the brain with minimal discomfort to patients, providing information about normal or abnormal brain-related conditions and providing decision-making support for physicians. The investigators hypothesize that the HS-1000 is capable of detecting vasospasm using the raw acoustic data derived from the noninvasive procedure.

DETAILED DESCRIPTION:
The study will be an open-label, non-randomized, prospective study in patients with elevated risk of vasospasm after stabilizing the patient and treating the subarachnoid hemorrhage (SAH) to prevent further re-bleeds.

Each enrolled patient will be monitored with the HS-1000 device for a period of 10 minutes, occurring daily, after completion of surgery for SAH. Following admittance to the intensive care unit (ICU), patients will undergo routine monitoring as per standard of care. Non-invasive recordings of 10 minutes in duration with HS-1000 device will be completed daily for up to 14 days contingent on staff availability and the patient's clinical status. In the event a monitoring session is interrupted or postponed, another attempt to re-monitor will be made when the patient is able. Flexibility will granted in lieu of patient or study team unavailability thereby allowing recording to be neglected for any given day if absolutely necessary.

In the case the principle investigator (PI) or a member of the study team positively confirms vasospasm based on clinical assessment or follow-up care of the patient during the monitoring period, the patient will be recorded twice daily for up to a consecutive 14 days or for their duration in the ICU. The PI will determine the severity of vasospasm as per the vasospasm severity scale. Increased recording frequency will be implemented only for patients with vasospasm graded as asymptomatic moderate-to-severe or symptomatic mild-to-severe (i.e. those scoring 2a, 3a, 1s, 2s, or 3s).

Prior to the HS-1000 recording session, the front-end will be placed in the patient's ears and connected to the monitor. The acoustic signal propagates through the cranium, and attenuates during its propagation. The receiving sensor in the other headset picks up the acoustic signal. The receiving sensor converts the acoustical signal into a digital signal and transmits it back to the monitor.

Each recording session with the HS-1000 will last 10 consecutive minutes, if the patient's condition and clinical workflow permits. If required by the attending medical staff, the recording can be stopped and restarted at a later time during the day. The HS-1000 will be used as a seamless adjunctive, state-of-the-art, brain monitoring utility operating in parallel with standard care intensive neurological monitoring modalities. The non-invasive monitor will not replace or alter the standard care received by patients. Once all recordings are completed, the brain monitoring signals will be saved in the study's database.

Daily neurological checks and collection of all routine clinical and radiographic data as per standard of care will be gathered as the gold standard data for statistical comparison. Neurocognitive tests will be performed routinely every 8 hours by attending physicians to assess for neuro-deterioration and radiological (Computed tomographic angiography (CTA) and Digital subtraction angiography (DSA) components. Data collected from patients will be stripped of all personal health identifiers. Each subject will receive a unique identifying patient number linking the individual to their deidentified clinical data set. Only the medical staff attending to the patient's standard care will be knowledgeable to the identity of the subject.

Once data is collected, results of the HS-1000 recording sessions will be analyzed and correlated with deidentified supporting clinical/radiological data to assist in the identification of vasospasm-specific acoustic waveform patterns.

Deidentified supporting clinical data will consist of standard care intensive neurological monitoring procedures currently used to confirm clinical diagnosis of vasospasm, principally based on evidence of neuro deterioration:

1. Computed tomographic angiography
2. Digital subtraction angiography
3. Neurocognitive clinical assessments
4. Routine clinical data as per standard of care

Study workflow and HS-1000 recording sessions will be fully compatible with and will not alter the standard of care received by the patients in any way.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women at least 18 years of age inclusive at the time of hospital admission for stabilization and treatment of the SAH
* Subjects receiving intensive care neurological monitoring per standard care following treatment of SAH
* Subject or legal authorized representative is able and willing to comply with the requirements of the protocol
* Subject or legal authorized representative is able to understand and sign written informed consent to participate in the study
* Subject is expected to undergo standard care neurological intensive monitoring for a maximum of 14 days
* Confirmed presence of a ruptured saccular aneurysm on angiography (catheter or CTA) and treated by neurosurgical clipping or endovascular coiling.
* Patient must have a modified Fisher of II to IV.
* The SAH should be between grades I-IV as defined by the World Federation of Neurological Surgery (WFNS).

Exclusion Criteria:

* Subject with ear disease, ear trauma
* Subjects with dural defects, punctures
* Subjects with severe head trauma in which the location and/or severity of the skull fracture(s), i.e. frank skull fracture or major joint dislocations may jeopardize HeadSense monitoring procedure
* Subjects with cerebral fluid (CSF) leakage from the ear (CSF Otorrhea)
* Reported allergy or hypersensitivity to any of the test materials or contraindication to test materials
* Subjects currently enrolled in or less than 30 days post-participation in other investigational device or drug study(s), or receiving other investigational agent(s)
* Any condition that may jeopardize study participation (e.g., abnormal clinical or laboratory finding) or interpretation of study results, or may impede the ability to obtain informed consent (e.g., mental condition)
* Patients who have a modified Fisher of 0 to I
* Patients who have a WFNS of V
* Presence of an intraventricular or intracerebral hemorrhage in absence of SAH or with only local, thin SAH
* Angiographic vasospasm prior to aneurysm repair procedure, as documented by catheter angiogram or CTA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The HS-1000 will measure intracranial pressure readings from the patient which will then be used to generate vasospasm-specific acoustic waveform patterns. | 14 days following SAH
  Development of vasospasm-specific acoustic waveform patterns
To compare the HS-1000 ability and accuracy in detecting vasospasm by measuring ICP values compared to other standard of care vasospasm diagnostic modalities such as DSA and CTA. | 14 days following SAH
  Detection of vasospasm
To determine HS-1000's ability and accuracy in measuring ICP values while assessing physiological parameters of the patient. | 14 days following SAH
  ICP measurement

SECONDARY OUTCOMES:
Incidence of Adverse events (AEs) | 48 hours from the end of monitoring with the HS-1000
  AE monitoring
Rate of ear infections/irritations | 48 hours from the end of monitoring with the HS-1000
  Side effects

OTHER OUTCOMES:
To evaluate the ergonomic and functional aspects of using the HS-1000 by having the operators of the device complete a brief 5 question survey about the ease or difficulty in using the device. | 2 months after data collection complete
  Function of the device

CONTACTS AND LOCATIONS:
Overall Officials: E. Francois Aldrich, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No